CLINICAL TRIAL: NCT03911089
Title: A Collection of Case Studies in Infants With Urea Cycle Disorders (UCD) to Evaluate Infant Growth and the Safety of a New Medical Food for UCD
Brief Title: A Collection of Case Studies in Infants With UCD to Evaluate Infant Growth and the Safety of a New Medical Food for UCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPR15IN89539
Record Dates: First submitted 2018-08-28; First posted 2019-04-10 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Urea Cycle Disorder; Inborn Errors of Metabolism
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label (Other): UCD Anamix Infant
  Interventions: Other: UCD Anamix Infant

INTERVENTIONS:
Other: UCD Anamix Infant — UCD Anamix infant with DHA and ARA is an amino acid based infant medical food containing only the essential amino acids, carbohydrate, fat, vitamins, minerals and trace elements.

SUMMARY:
Original study: Study aims to enroll 3-5 children with confirmed Urinary Cycle Disorder (UCD). Subjects meeting the inclusion and exclusion criteria are included during the baseline visit. All subjects will receive the investigational product for a period of 16 weeks. At baseline, 2, 4, 8, 12 and 16 weeks the study parameters are assessed.

The study amendment aims to collect case studies retrospectively of children who have used UCD Anamix Infant for at least 16 weeks, in countries where UCD Anamix Infant is already available on the market. It is aimed to collect the same study parameters of the original study at preferably the same timepoints.

ELIGIBILITY:
Inclusion criteria:

Prospective study:

* Male and female infants diagnosed with UCD, aged from birth to 30 days of age
* Parent / primary caregiver is able to give informed consent
* Infants who will receive and will be able to take study medical food as part (40-70%) of their protein requirements in the day

Retrospective study:

* Male and female term infants diagnosed with UCD, that started UCD Anamix Infant when aged from birth to 30 days of age.
* Parent / primary caregiver is able to give informed consent
* Infants who received UCD Anamix Infant as part of their protein requirements (40-70%) in the day for at least 16 weeks.

Exclusion Criteria:

* Infants < 5lb 8oz (< 2.5 kg) at birth
* Infants <34 weeks of gestation and using a special premature formula at study start
* Infants with severe concurrent illness or major congenital malformations, except conditions consequent to urea cycle disorder
* Infants with suspected or documented systemic or congenital infections (e.g. human immunodeficiency virus)
* Infants with evidence of significant cardiac, respiratory, haematological, gastrointestinal, or other systemic diseases
* Infants currently taking cytotoxic drugs
* Investigator's uncertainty about the willingness or ability of the parent to comply with the protocol requirements
* Participation in any other study involving investigational products concomitantly or prior to entry into the study
* An infant of any personnel connected with the study
* Infants whose parent / primary caregiver is younger than the legal age of consent

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2013-05-28 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Growth: weight | 16 weeks
  weight [kg]
Growth: length | 16 weeks
  length [cm]
Growth: head circumference | 16 weeks
  head circumference [cm]

SECONDARY OUTCOMES:
GI symptoms [absent/mild/moderate/severe] | 16 weeks
  GI symptoms for the following symptoms:
  * Vomiting (>1 tablespoon/15ml)
  * Abdominal distension
  * Burping
  * Flatulence
  * Diarrhoa
  * Constipation
  * Colic (cramps)
  * Regurgitation (<1 tablespoon/15ml)
Stool frequency | 16 weeks
  stool frequency [# times/day]
Stool consistency | 16 weeks
  stool consistency: quantification score: [Watery; Soft, puddinglike; Soft, formed; Dry, formed; Dry, hard pellets]
Compliance: product intake | 16 weeks
  Intake of medical food compared to amount prescribed [ volume: ml per day]
Protein and iron levels from blood samples (for retrospective study part only if data available) | 16 weeks
  Protein, amino acids and nutrient levels in blood [g/dL] or [umol/L]

OTHER OUTCOMES:
Safety and tolerability: (S)AE | 16 weeks
  Occurence of (Serious) Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Philadelphia, Philadelphia, Pennsylvania, United States